CLINICAL TRIAL: NCT02489214
Title: A Phase 1B Study of Donafenib Monotherapy for Previously Treated Metastatic Gastric Cancer
Brief Title: Donafenib Monotherapy for Previously Treated Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate policy adjustments
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGDG1B
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer
Keywords: donafenib
MeSH Terms: conditions — Stomach Neoplasms | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- donafenib tosilate tablets (Experimental): 200mg bid
  Interventions: Drug: donafenib tosilate tablets

INTERVENTIONS:
Drug: donafenib tosilate tablets — 200mg bid
  Other Names: CM4307

SUMMARY:
This open-label, one-center, noncomparative, two-stage phase 1B trial assessed the donafenib in advanced gastric cancer.

DETAILED DESCRIPTION:
This open-label, one-center, noncomparative, two-stage phase 1B trial assessed the tyrosine kinase inhibitor donafenib tosilate tablets (400 mg/d,200mg bid) in patients with advanced, inoperable gastric cancer progressing after chemotherapy . The primary endpoint is the safety.The secondary endpoints are tumor response and progression-free survival time.

ELIGIBILITY:
Inclusion Criteria:

* All patients provided written, informed consent.
* Have histological or cytological documentation of gastric adenocarcinoma;
* Have received currently approved standard therapies and to have disease progression during or within 3 months after the last administration of the last standard therapy or to have stopped standard therapy because of unacceptable toxic effects.
* Standard therapies include as many of the following as were licensed: a fluoropyrimidine,oxaliplatin,irinotecan, paclitaxel,docetaxel;and trastuzumab for patients who had Her-2 positive tumours;
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Life expectancy of at least 3 months;
* Have adequate bone-marrow, liver, and renal function at the start of the trial.
* Prothrombin time international normalized ratio≤1.5；

Exclusion Criteria:

* Patients with brain metastases.
* Patients receiving cytotoxic chemotherapy, immunotherapy or hormonal therapy, radiotherapy to site of measurable or evaluable disease within the previous 4 weeks.
* Patients had evidence of clinically active interstitial lung disease or abnormal blood results by predefined criteria (serum bilirubin >1.5 times upper limit of reference range, aspartate or alanine aminotransferase>2.5 times the upper limit of normal if no demonstrable liver disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 54 weeks
  patients with adverse events/all patients*100%

SECONDARY OUTCOMES:
Tumor response | 54 weeks
  complete response and partial response patients/all patients*100%
Progression-free survival time | 54 weeks
  median progress-free survival time

CONTACTS AND LOCATIONS:
Overall Officials: Bao Rui, Doctor, Principal Investigator — The affiliated hospital of Nanjing University Medical School
Locations (2):
- China (2):
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Affiliated Cancer Center of Academy of Military Medical Sciences, Beijing